CLINICAL TRIAL: NCT01970566
Title: Effect of Intense-Exercise/Moderate-Calorie vs Topiramate-Phentermine on Obesity
Brief Title: Comparison of the Effect of Intense-Exercise/Moderate-Calorie, Topiramate-Phentermine and Cognitive Behavioral Therapy on Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The project was not announced to the field and it was not funded.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-001-12F
Record Dates: First submitted 2013-08-28; First posted 2013-10-28 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Obesity; Diabetes Mellitus
Keywords: Intense Exercise/Moderate Calorie Restriction; Topiramate-Phentermine
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IE-MCR (Experimental): Intense Exercise/Moderate Calorie Restriction
  Interventions: Other: Behavioral
- TP-CBT (Active Comparator): Topiramate-Phentermine plus cognitive behavioral therapy
  Interventions: Other: Behavioral and Drug
- CBT (Active Comparator): cognitive behavioral therapy
  Interventions: Other: Behavioral and Drug; Other: Behavioral

INTERVENTIONS:
Other: Behavioral and Drug — Topiramate-Phentermine plus cognitive behavioral therapy
  Other Names: TP-CBT
  Arms: TP-CBT
Other: Behavioral — Intense Exercise/Moderate Calorie Restriction
  Other Names: IE-MCR
  Arms: IE-MCR
Other: Behavioral and Drug — Topiramate-Phentermine plus cognitive behavioral therapy
  Other Names: TP-CBT
  Arms: CBT
Other: Behavioral — Intense Exercise/Moderate Calorie Restriction
  Other Names: IE-MCR
  Arms: CBT

SUMMARY:
Obesity is a prevalent disorder and linked with inflammation, insulin resistance, dyslipidemia, obstructive sleep apnea, atherosclerosis, and associated with significant morbidity and mortality. This randomized clinical trial will compare the effectiveness of Intense Exercise/Moderate Calorie Restriction (IE-MCR), Topiramate-Phentermine (TP) and cognitive behavioral therapy (CBT) on obesity and atherosclerosis in individuals with morbidly obesity. This randomized clinical trial will compare: 1) the change in fat mass and atherosclerosis, 2) the change in psychological and quality-of-life as well as economic burden in response to IE-MCR, TP and CBT, and 3) conduct exploratory mechanistic biomolecular, genetic and therapeutic analyses to develop intervention-specific individualized intervention models to improve management of morbidly obese individuals.

DETAILED DESCRIPTION:
Background. Obesity is prevalent disorder; up to 60% of US population that is associated with significant morbidity and mortality through inflammation, insulin resistance, dyslipidemia, obstructive sleep apnea, and atherosclerosis. The economic burden of obesity-related illnesses is substantial, with estimates ranging from 2% to 7% of the total US health care expenditures and billions of dollars in direct and indirect costs to society. This randomized clinical trial will compared the effectiveness of Intense Exercise/Moderate Calorie Restriction (IE-MCR), Topiramate-Phentermine (TP) and cognitive behavioral therapy (CBT) on obesity and atherosclerosis in morbidly obesity individuals (body mass index(BMI)>40 kg/m2 or BMI>35 kg/m2 with associated comorbidities) with diabetes mellitus (DM).

Importance/Significance. There is a cumulative increase in the rate of obesity, up to 60% of the US population. This randomized clinical trial will compare: 1) the change in fat mass and atherosclerosis and, 2) the change in psychological status and quality-of-life as well as economic burden in response to IE-MCR, TP and CBT in morbidly obese individuals with DM. Furthermore, 3) exploratory analyses evaluating the different underling adipocyte molecular mechanisms will be conducted. This will investigate the underlying genomic determinants and characterizes the management of obesity by comparing biologic, clinical phenotype, and cost effectiveness of these two interventions. These aims will provide fundamental information to assess the beneficial effects within and across interventions on obesity and atherosclerosis management which will help provide individualized intervention models to improve management of morbidly obese individuals Method. A significant difference in reduction of fat mass, carotid/coronary atherosclerosis, improve in psychological, quality of life and economic burden measures, as well as exploratory mechanism of action across IE-MCR, TP and CBT methods, are hypothesized. Over a 5 year period, 60 morbidly obese individuals with diabetes mellitus aged 18 or older and free of clinical cardiovascular disease will be recruited from the Obesity Clinic of the Greater Los Angeles VA Health Care System, University of California Los Angeles and Captain Lovell Federal Healthcare Center. Eligible subjects will be randomized to either of intense exercise/moderate calorie restriction, Topiramate-Phentermine or cognitive behavioral therapy (20 in each group) and receive these intervention for 12-months. Intense exercise/moderate calorie restriction group will receive lectures on exercise and general dietary measures including calorie counting. They will prepare their own food, with protein:carbohydrate:fat ratio of 30:45:25 and over 70% of their resting daily energy expenditure (RDEE), and completed daily food and exercise journals. They will exercise ~2.5 hours/day, about 1/4 supervised, for a year. Topiramate-Phentermine group will receive full dose of TP (15/92mg) pills daily for a period of 1-year. Furthermore, CBT group as well as IE-MCR and TP will receive weekly cognitive behavior therapy for a year. All subjects will undergo carotid ultrasound; coronary computed tomography angiography, bioelectric impedance spectroscopy, dual-energy X-ray absorptiometry, ambulatory calorimetry, serial home resting metabolic rate serial home (RMR),sleep apnea assessment and abdominal fat pad fine-needle aspiration biopsy (FNAB), as well as measurement of oxidative stress/inflammatory/metabolic biomarkers at baseline and at 1-year follow-up. Quality of life, psychological health and economic burden will be assessed using standardized questionnaires. Participants will complete quarterly trial visits for physical exam, compliance to intervention as well as ascertainment of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70 years
* Competent to give informed consent
* Obesity (BMI>40) or BMI>35 kg/m2 with associated co-morbidities
* Diabetes Mellitus Type II

Exclusion Criteria:

* History of coronary artery disease, myocardial infarction, coronary angioplasty or bypass surgery
* Prior non-cardiac illness with an estimated life expectancy <4 years
* Unable to give informed consent
* Women who are pregnant or lactating
* Prior bariatric surgery or receiving anti-obesity drugs

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Compare the rate of change in fat mass in intense exercise/moderate diet restriction, topiramate-phentermine and cognitive behavior therapy | 12 month and 24 month Follow Ups
  compare the change in extracellular/total body water, body fat/lean mass and metabolically active adipose tissue in response to IE-MCR vs. TP-CBT.

SECONDARY OUTCOMES:
Compare the rate of atherosclerotic burden in intense exercise/moderate diet restriction, topiramate-phentermine and cognitive behavior therapy | 12 month and 24 month Follow Ups
  Compare the change in carotid intima media thickness, coronary artery distensibility index and plaque volume in response to IE-MCR,TP or CBT.
Compare the change in neuropsychiatric status in response to intense exercise/moderate diet restriction, topiramate-phentermine and cognitive behavioral therapy | 12 month and 24 month Follow Ups
  compare the change in cognition, anxiety, depression and vitality in response to IE-MCR, TP and CBT.
Comparison the rate of and atherosclerotic burden in intense exercise/moderate diet restriction, topiramate-phentermine and cognitive behavior therapy | 12 month and 24 month Follow Ups
  Compare the change in carotid intima media thickness, coronary artery distensibility index and plaque volume in response to IE-MCR,TP or CBT.
Compare the change in quality-of-life in response to intense exercise/moderate diet restriction, topiramate-phentermine and cognitive behavioral therapy | 12 month and 24 month Follow Ups
  Compare the change in satisfaction, well-Being and quality of life in response to IE-MCR, TP and CBT

CONTACTS AND LOCATIONS:
Overall Officials: Naser Ahmadi, MD MS PhD, Principal Investigator — Captain James A. Lovell Federal Health Care Center, North Chicago, IL
Locations (1):
- Captain James A. Lovell Federal Health Care Center, North Chicago, IL, North Chicago, Illinois, United States

REFERENCES:
- [Background] Ahmadi N, Tsimikas S, Hajsadeghi F, Saeed A, Nabavi V, Bevinal MA, Kadakia J, Flores F, Ebrahimi R, Budoff MJ. Relation of oxidative biomarkers, vascular dysfunction, and progression of coronary artery calcium. Am J Cardiol. 2010 Feb 15;105(4):459-66. doi: 10.1016/j.amjcard.2009.09.052. PMID 20152239
- [Result] Ahmadi N, Eshaghian S, Huizenga R, Sosnin K, Ebrahimi R, Siegel R. Effects of intense exercise and moderate caloric restriction on cardiovascular risk factors and inflammation. Am J Med. 2011 Oct;124(10):978-82. doi: 10.1016/j.amjmed.2011.02.032. Epub 2011 Jul 27. PMID 21798505